CLINICAL TRIAL: NCT01736436
Title: APG101 in Transfusion-Dependent Patients With Low or Intermediate Risk Myelodysplastic Syndrome
Brief Title: APG101 in Myelodysplastic Syndrome
Acronym: APG101 in MDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Apogenix GmbH (Industry)
Responsible Party: Sponsor
Organization: Apogenix AG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APG101_CD_003; 2012-003027-37 (EudraCT Number)
Record Dates: First submitted 2012-11-14; First posted 2012-11-29 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Myelodysplastic Syndrome
Keywords: MDS; Myelodysplastic syndrome; Low and intermediate risk; Transfusion-dependent patients; Transfusion; Anemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — Therapeutics; APG101

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 100 mg APG101 weekly over 12 weeks (Experimental): Single arm open label study. Patient receive 100 mg APG101 i.v. weekly over 12 weeks with a 6 monthly follow-up phase
  Interventions: Drug: Treatment with APG101; Procedure: Bone marrow collection; Procedure: Blood drawings

INTERVENTIONS:
Drug: Treatment with APG101 — Patients will be treated 12 weeks with 100 mg APG101 intravenous weekly
Procedure: Bone marrow collection — During the study, bone marrow will be collected 4 times to assess study objectives
Procedure: Blood drawings — During the study, blood will be drawn at different time points to assess study objectives

SUMMARY:
It has been shown in preclinical experiments with bone marrow from patients with myelodysplastic syndrome that APG101 rescues erythrocytes from premature cell death. This is expected to translate in an improved erythropoiesis and ameliorated anemia in MDS patients.

APG101 might, therefore, be a valuable addition to current treatments of low- or intermediate MDS patients suffering from anaemia.

Transfusion-dependent patients with low or intermediate risk MDS according to WHO Prognostic Scoring Scale (WPSS) can be included in this study.

Treatment consists of 100mg APG101 intravenous as a weekly treatment over 12 weeks + 6 months follow up phase.

Primary objective of the trial is safety and tolerability of APG101; secondary objectives are

* Hematologic, cytologic and cytogenetic response rate using modified International Working Group (IWG) response criteria
* Incidence and time to leukemic progression at 37 weeks
* OS (Overall survival) at 37 weeks

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male and female patients with cytologically or histologically established diagnosis of de novo MDS according to the WHO-classification, either previously treated or untreated, presenting with low or intermediate risk features according to WHO prognostic status scale (WPSS)
* Diagnosis of MDS with a medullary blast count of less than 5% has to be established or confirmed by bone marrow morphology
* MDS with 5q deletion only if Lenalidomide is not a treatment option
* Red blood cell transfusion dependency of at least 4 units of packed red blood cells (PRBC) during the last 8 weeks before inclusion. Only PRBC transfusions given for a Hb level ≤ 9g/dl or a haemoglobin level > 9g/dl, if clinically indicated (e.g. coronary heart disease, long distance travel), will count.
* Patients refractory to Erythropoietin-stimulating agents (ESA) (as assessed after at least 8 weeks of treatment) or with a low possibility to respond to ESA treatment
* at least 18 years old, smoking or non-smoking, of any ethnic origin
* ECOG performance status ≤ 2
* Suitable veins or existing port system for intra-venous infusion
* Adequate contraception

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* MDS with medullary blast count ≥ 5%
* Chronic monomyeloic leucemia (CMML)
* Therapy-related / secondary MDS
* High-risk karyotype according to WPSS
* Patients scheduled for bone marrow or stem cell transplant within the next 6 months
* Parallel treatment with ESA or with other experimental therapy
* Prior chemotherapy (including Vidaza)
* Treatment within the last 6 weeks with histone deacetylase (HDAC) inhibitors or ESAs
* Treatment within any other clinical trial parallel to the treatment phase of the current study or within 30 days before inclusion
* Active uncontrolled infection
* HIV, active hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection
* Any other condition / treatment or past medical history of diseases with poor prognosis that, in the opinion of the investigator, might interfere with the study
* History of or current drug or substance abuse
* History of other (haemato-) oncological disease (except for non-melanoma skin cancer and adequately treated in situ carcinoma of the cervix)
* Inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study
* Unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study
* Subject is the investigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study.
* Hypersensitivity to recombinant proteins or excipients in the investigational drug
* Pregnancy or breast feeding
* Vulnerable patients (e.g., minors or persons kept in detention)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | During the whole study (37 weeks)
  Evaluation of adverse events (AEs) and serious adverse events (SAEs). Evaluation of electrocardiograms (ECGs), abdominal ultrasound, anti-drug antibodies (ADA), changes in lymphocyte subpopulations / activation markers and changes in performance status (ECOG).
  Any side effects potentially related to the APG101 treatment are evaluated.

SECONDARY OUTCOMES:
Overall survival (OS) | OS is captured for 37 weeks (during study)
  Overall survival (OS) is defined as time from start of study treatment to death from any cause
Changes in transfusion frequency | During the whole study. Baseline values are compared to values under treatment with APG101 (e.g baseline compared to week 12 and week 37)
  Changes in transfusion frequency will be evaluated as those are early signs of an improval in erythropoiesis
Changes of different parameters (e.g. histologic, cytologic, cytogenetic) in bone marrow according to Chesson criteria | During the study (37 weeks)
  By assessing different parameters (cytologic, hematologic, cytogenetic), safety as well as efficacy of treatment with APG101 can be evaluated
Changes in hemoglobin (Hb) level | During the study (37 weeks)
  Changes in Hb level will be evaluated as those are early signs of an improval in erythropoiesis

CONTACTS AND LOCATIONS:
Overall Officials: Florian Nolte, MD, Principal Investigator — Universitaetsmedizin Mannheim, III. Medizinische Klinik, Hämatologie und Onkologie, Theodor-Kutzer-Ufer 1-3, 68167 Mannheim, Germany
Locations (2):
- Germany (2):
  - Universitaetsklinik Heidelberg, Medizinische Klinik V, Haematologie, Onkologie & Rheumatologie, Heidelberg
  - Universitaetsmedizin Mannheim, III. Medizinische Klinik, Haematologie und Onkologie, Mannheim